CLINICAL TRIAL: NCT03540147
Title: The Impact of Blood Flow Restriction (BFR) on Exercise and Hemodynamic Responses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of subjects in this study was overestimated in the initial assessment.
Sponsor: University of Texas at Austin (Other)
Collaborators: Savannah Wooten (Unknown); Stray-Gundersen, Sten, Ph.D. (Individual)
Responsible Party: Principal Investigator, Hirofumi Tanaka, Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-10-0074
Record Dates: First submitted 2018-04-30; First posted 2018-05-30 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Exercise Training; Hemodynamic Response
Keywords: blood flow restriction; blood pressure; yoga

STUDY DESIGN:
Intervention Model Description: Each participant will undergo five visits to the laboratory for repeated testing under five different conditions. The sessions will be randomized and will take 2.5 hours to complete.
Who Masked: Participant
Masking Description: The participants will not know which condition they will receive on the day of testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Exercise with Hokanson cuffs (Experimental): Participants will walk on the treadmill with Hokanson cuffs inflated.
  Interventions: Device: Hokanson Cuffs
- Exercise with BStrong Bands (Experimental): Participants will walk on the treadmill with BStrong bands inflated.
  Interventions: Device: BStrong Bands
- Exercise without inflated bands/cuffs (Sham Comparator): Participants will walk on the treadmill with non-inflated BStrong bands.
  Interventions: Device: BStrong Bands
- Yoga poses with BStrong bands inflated (Experimental): Participants will perform 15-20 yoga poses with BStrong bands inflated.
  Interventions: Device: BStrong Bands
- Yoga poses with BStrong bands uninflated (Sham Comparator): Participants will perform 15-20 yoga poses with uninflated BStrong bands.
  Interventions: Device: BStrong Bands

INTERVENTIONS:
Device: Hokanson Cuffs — Each subject will participate in all (5) experimental arms. The order in which the experimental arms will be completed will be randomly assigned to the participant.
  Arms: Exercise with Hokanson cuffs
Device: BStrong Bands — Each subject will participate in all (5) experimental arms. The order in which the experimental arms will completed will be randomly assigned to the participant.
  Arms: Exercise with BStrong Bands; Exercise without inflated bands/cuffs; Yoga poses with BStrong bands inflated; Yoga poses with BStrong bands uninflated

SUMMARY:
The impact of blood flow restriction (BFR) on exercise and hemodynamic responses will be studied. The use of BFR will be studied during yoga and low-intensity aerobic exercise in healthy subjects with no history of chronic illness ranging from 18-40 years of age. This study will evaluate several conditions related to cardiovascular physiology in order to determine the safety and efficacy of this type of exercise training. First, the effects of two distinct types of BFR cuffs (BStrong and Hokanson) will be studied during low-intensity aerobic exercise on vascular function. Second, the effect of yoga will be studied with and without the use of BStrong bands on vascular function. Outcome measures include acute effects on endothelial function i.e. flow-mediated dilation, arterial stiffness, beat-by-beat blood pressure, heart rate, RPE (rate of perceived exertion), and blood lactate. For this intervention, the BFR cuffs will be used during exercise to evaluate its safety and efficacy. Since BFR is becoming a widely popular method of exercise, it is important to study its safety and hemodynamic effects.

DETAILED DESCRIPTION:
Participants will be tested a total of 5 times; twice for the yoga portion and thrice for the aerobic exercise (walking) portion. Outcome measures will be consistent across the five visits and will take approximately 2.5 hours to complete. The order of the five separate sessions will be randomized such that the participant cannot expect which condition they will be performing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Pregnancy
* A recent illness, recent surgery, or any medical intervention
* history of diabetes, heart disease, or other cardiovascular problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2019-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Tanaka, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Cardiovascular Aging Research Lab at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD without identifying information will be shared with other investigators with a reasonable request to the investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The information is available now.
Access Criteria: They will be available with a reasonable request to the investigators.

REFERENCES:
- [Background] Renzi CP, Tanaka H, Sugawara J. Effects of leg blood flow restriction during walking on cardiovascular function. Med Sci Sports Exerc. 2010 Apr;42(4):726-32. doi: 10.1249/MSS.0b013e3181bdb454. PMID 19952840
- [Background] Sugawara J, Tomoto T, Tanaka H. Impact of leg blood flow restriction during walking on central arterial hemodynamics. Am J Physiol Regul Integr Comp Physiol. 2015 Oct;309(7):R732-9. doi: 10.1152/ajpregu.00095.2015. Epub 2015 Aug 5. PMID 26246503
- [Background] Shimizu R, Hotta K, Yamamoto S, Matsumoto T, Kamiya K, Kato M, Hamazaki N, Kamekawa D, Akiyama A, Kamada Y, Tanaka S, Masuda T. Low-intensity resistance training with blood flow restriction improves vascular endothelial function and peripheral blood circulation in healthy elderly people. Eur J Appl Physiol. 2016 Apr;116(4):749-57. doi: 10.1007/s00421-016-3328-8. Epub 2016 Jan 28. PMID 26822582
- [Background] Hunter SD, Dhindsa MS, Cunningham E, Tarumi T, Alkatan M, Nualnim N, Tanaka H. The effect of Bikram yoga on arterial stiffness in young and older adults. J Altern Complement Med. 2013 Dec;19(12):930-4. doi: 10.1089/acm.2012.0709. Epub 2013 Jun 5. PMID 23738677
- [Background] Miles SC, Chun-Chung C, Hsin-Fu L, Hunter SD, Dhindsa M, Nualnim N, Tanaka H. Arterial blood pressure and cardiovascular responses to yoga practice. Altern Ther Health Med. 2013 Jan-Feb;19(1):38-45. PMID 23341425
- [Background] Hunter SD, Dhindsa MS, Cunningham E, Tarumi T, Alkatan M, Nualnim N, Tanaka H. Impact of Hot Yoga on Arterial Stiffness and Quality of Life in Normal and Overweight/Obese Adults. J Phys Act Health. 2016 Dec;13(12):1360-1363. doi: 10.1123/jpah.2016-0170. Epub 2016 Aug 24. PMID 27633625
- [Derived] Stray-Gundersen S, Wooten S, Tanaka H. Walking With Leg Blood Flow Restriction: Wide-Rigid Cuffs vs. Narrow-Elastic Bands. Front Physiol. 2020 May 29;11:568. doi: 10.3389/fphys.2020.00568. eCollection 2020. PMID 32547424

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross-over study. Each subject performed all 5 experimental conditions that includes "exercise with Hokanson cuffs", "Exercise with BStrong bands", "Exercise without inflated bands/cuffs", "Yoga poses with BStrong bands inflated" and "Yoga poses with BStrong bands uninflated". The number of subjects studied is 20.
Groups:
- Blood Flow Restriction Exercise: This is a cross-over study. Each subject performed all 5 experimental conditions that includes "exercise with Hokanson cuffs", "Exercise with BStrong bands", "Exercise without inflated bands/cuffs", "Yoga poses with BStrong bands inflated" and "Yoga poses with BStrong bands uninflated".
Period: Overall Study
Arm/Group | Blood Flow Restriction Exercise
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Blood Flow Restriction Exercise: Participants will walk on the treadmill with Hokanson cuffs inflated.
  Hokanson Cuffs: Each subject will participate in all (5) experimental arms. The order in which the experimental arms will be completed will be randomly assigned to the participant.
Arm/Group | Blood Flow Restriction Exercise
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 23 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body weight [Mean (Standard Deviation); unit: kg] | 71 (10)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Arterial blood pressure was measured using the automatic oscillometric methods.
Time Frame: Measurements were taken at Baseline (before Experimental Arm Participation) and immediately after Experimental Arm Participation.
Population: Baseline (before Experimental Arm Participation) data are reported below.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exercise With Hokanson Cuffs | Exercise With BStrong Bands | Exercise Without Inflated Bands/Cuffs | Yoga Poses With BStrong Bands Inflated | Yoga Poses With BStrong Bands Uninflated
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
mmHg
  Baseline (before the experimental arm participation) | 116 (11) | 116 (9) | 117 (7) | 117 (7) | 115 (8)
  Immediately after | 150 (16) | 127 (10) | 158 (14) | 160 (15) | 130 (15)

2. Primary Outcome: Flow-mediated Dilation
Description: After 20 minutes of supine rest, endothelial function was measured via flow-mediated dilation (FMD) technique by measuring the brachial artery's diameter increase following a brief period of occlusion using an automated diagnostic ultrasound system. A blood pressure cuff was placed on the forearm with the proximal edge of the cuff above with the participant's antecubital fossa. Two cross-sectional images of the artery were acquired utilizing the automated ultrasound probe proximal to the antecubital fossa. Following baseline metrics, the cuff was inflated to 50 mmHg above resting systolic blood pressure for 5 minutes to occlude blood flow. After 5 minutes of occlusion, the cuff was deflated, and both brachial artery diameter and blood flow velocity were measured simultaneously and continuously for two-minutes immediately post occlusion. FMD was calculated as a percent increase in brachial artery diameter at the post-blood flow occlusion compared with the pre-blood flow occlusion.
Time Frame: Before (baseline) and after the exercise interventions
Measure: Mean (Standard Error); unit: percentage of resting diameter
Arm/Group | Exercise With Hokanson Cuffs | Exercise With BStrong Bands | Exercise Without Inflated Bands/Cuffs | Yoga Poses With BStrong Bands Inflated | Yoga Poses With BStrong Bands Uninflated
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
percentage of resting diameter
  Baseline (before conditions) | 7.0 (2) | 7.2 (2.2) | 7.0 (1.8) | 6.8 (1.6) | 6.9 (2)
  After conditions | 6.8 (1.8) | 7.1 (2.0) | 7.1 (1.9) | 7.0 (2) | 6.7 (1.7)

ADVERSE EVENTS:
Time Frame: Each participants came to the laboratory twice in the span of 2 weeks.
Arm/Group | Exercise With Hokanson Cuffs | Exercise With BStrong Bands | Exercise Without Inflated Bands/Cuffs | Yoga Poses With BStrong Bands Inflated | Yoga Poses With BStrong Bands Uninflated
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03540147/Prot_SAP_001.pdf